CLINICAL TRIAL: NCT04181645
Title: SHR- 1210 Combined With Paclitaxel (Albumin Bound) and Gemcitabine as First-line Therapy in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPOG1210-003
Record Dates: First submitted 2019-11-25; First posted 2019-11-29 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer Stage IV
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to accept the combination treatment of SHR-120 with Paclitaxel-albumin and gemcitabine after meeting the inclusion criteria.
Masking Description: An open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-120, Paclitaxel-albumin and Gemcitabine (Experimental): Subjects receive SHR-1210 200mg (Day 1) and Paclitaxel-albumin 125mg/m2 (Day1 and Day8) and gemcitabine 1000mg/m2 (Day 1 and Day 8) of each 21-day cycle for at most 6 cycles until documented PD or intolerable adverse event or new anti-cancer treatment or loss to follow-up or death.
  Subjects receive SHR-1210 200mg (Day1) to maintain after 6 cycles treatment without PD or listed situation to terminate.
  Interventions: Drug: Biological: SHR-1210 Drug: Gemcitabine Drug:Paclitaxel-albumin

INTERVENTIONS:
Drug: Biological: SHR-1210 Drug: Gemcitabine Drug:Paclitaxel-albumin — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody. Gemcitabine Other Name: Gemcitabine Hydrochloride for Injection Paclitaxel-albumin Other Name: Paclitaxel-albumin Injection

SUMMARY:
This is an open-label, single center, non-randomized, phase I trial to evaluate safety and efficacy of using the combination treatment of SHR-1210 with Paclitaxel-albumin and gemcitabine of metastatic PDAC.

DETAILED DESCRIPTION:
This is an open-label, single center, non-randomized, phase I trial to evaluate safety and efficacy of using the combination treatment of SHR-1210 with Paclitaxel-albumin and gemcitabine of metastatic PDAC.

PD-1 antibody SHR-1210 is a humanized monoclonal antibody, and the heavy chain is immunoglobulin G4 (IgG4), the light chain is immunoglobulin κ (IgK). SHR-1210 specifically binds to PD-1 and blocks the interaction of PD-1 with its ligand (PD-L1), allowing T cells to recover against tumor immune responses.

The safety of SHR-1210 will be assessed by ongoing reviews of clinical laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status, physical examination, electrocardiogram (ECG), and adverse events. Evaluations of immune safety will also be conducted (immune-related adverse events (AEs), or labs of autoimmune sera, inflammatory events, and immunogenicity). Safety evaluations (both clinical and laboratory) are performed at baseline, before each study treatment, and throughout the study.

Tumor response will be assessed by radiographic examination in screening visit and every 2 cycles after first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >= 18 years, male or female;
2. Histologically or Cytologically confirmed metastatic pancreatic adenocarcinoma;
3. Patients have never received systematical anti-cancer therapy;
4. Based on Response Evaluation Criteria In Solid Tumors (RECIST1.1), there should be at least one measurable lesion which has never received local treatment like radiotherapy(The lesion located in previous radiotherapy areas can also be selected as target lesions if the progress confirmed.)
5. ECOG:0-1;
6. Expected survival>=12 weeks;
7. Essential organs function must meet the following criteria (Any blood products, growth factor, leucocyte promoting drugs, platelet promoting drugs, drugs for anemia are not allowed in 14 days before the first use of the experimental medication):

1) Absolute neutrophil count(ANC) >= 1.5x10^9/L 2) Platelet >= 85x10^9/L 3) Hemoglobin >= 90g/L 4) Serum Albumin >= 30g/L 5) Total bilirubin <= 2.0 ULN (Biliary obstructive patients after biliary drainage <= 2.5 ULN), AST and ALT <= 3.0 ULN (patients with liver metastasis <= 5 ULN); 6) Creatinine clearance rate >60 mL/min; 7) Activated Partial Thromboplastin Time and International Standardized Ratio <= 1.5 ULN (Patients using stable dose of anticoagulant therapy such as low molecular weight heparin or warfarin and INR is within the expected range of anticoagulants can be selected.)

Exclusion Criteria:

1. Patients with central nervous system metastasis.
2. Patients only have local advanced diseases.
3. Patients have uncontrolled pleural, pericardial or abdominal effusion requiring drainage.
4. Patients with history of allergy to monoclonal antibodies, any component of SHR-1210, paclitaxel(Albumin Bound) and Gemcitabine.
5. Patients have ever received anti PD-1 or anti PD-L1 therapy in the past.
6. Patients have accepted any experimental medication.within 4 weeks before the first dose of our experimental medication administration.
7. Patients are enrolled in another clinical trial except for observational clinical trial (Non-interventional) or the follow-up of the interventional clinical trial.
8. Patients accepted the last dose of anti-cancer therapy (including radiotherapy) within 4 weeks before the first dose of experimental medication administration.
9. Patients who need corticosteroid or other immunosuppressive agents.
10. Patients who ever received anti-cancer vaccine or have received live vaccine within 4 weeks before the first dose of administration.
11. Patients who have received major surgery within 4 weeks before the first dose of administration.
12. Patients with active autoimmune diseases, history of autoimmune diseases.
13. History of immunodeficiency, including HIV positive test, or other acquired, congenital immunodeficiency disorders, or history of organ transplantation and allogeneic bone marrow transplantation.
14. Patients with uncontrolled cardiovascular clinical symptoms or diseases.
15. Severe infections occurred within 4 weeks before the first administration.
16. History of interstitial lung disease and non- infectious pneumonia.
17. Patients with active pulmonary tuberculosis (APTB) infection confirmed by medical history or CT examination.
18. Patients with active hepatitis B or hepatitis C.
19. Patients with any other malignant tumors diagnosed within 5 years before the first administration.
20. Pregnant or lactating women.
21. According to the researchers, participants have other factors that may force them to end up the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
ORR：Objective Response Rate by IRC | through study completion, an average of 2 year
  objective response rate evaluated by Independent Review Committee using radiographic examination according to RECIST1.1

SECONDARY OUTCOMES:
ORR：Objective Response Rate by investigator | through study completion, an average of 2 year
  objective response rate evaluated by investigator using radiographic examination according to RECIST1.1
DCR: disease control rate | through study completion, an average of 2 year
  partial rate of subjects evaluated as CR/PR/SD in all subjects
DoR：duration of response | through study completion, an average of 2 year
  time firstly evaluated as CR or PR to time firstly evaluated as PD
PFS: progression-free survival | through study completion, an average of 2 year
  time from randomization to progression
OS: overall survival | through study completion, an average of 2 year
  time from randomization to death

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Wang, MD, Principal Investigator — RenJi Hospital
Locations (1):
- RenJiH, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jiujie Cui, Haiyan Yang, Jiong Hu, Jiayu Yao, Yu Wang, Yiyi Liang, Yongchao Wang, Feng Jiao, Xiaofei Zhang, Xiao Zhang, Ting Han, Tiebo Mao, Qing Xia, Xiuying Xiao, Li-Wei Wang. Anti-PD-1 antibody combined with albumin-bound paclitaxel and gemcitabine (AG) as first-line therapy and Anti-PD-1 monotherapy as maintenance in metastatic pancreatic ductal adenocarcinoma (PDAC). J Clin Oncol 39, 2021 (suppl 15; ASCO2021 abstr e16218).